CLINICAL TRIAL: NCT01456624
Title: A Randomized, Open Label, Single Dose, Cross-over, Phase I Trial to Investigate Safety and Pharmacokinetics of DW-ES(B) and Megace® Under Fasting and Fed Conditions in Healthy Male Volunteers
Brief Title: Phase 1 Study of Daewon-ES(B) & Megace in Healthy Male Volunteers Under Fasting and Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Gyu-Jeong Noh, Professor, Asan Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-0686
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Megace / Fasting condition (Active Comparator): 800mg
  Interventions: Drug: Megace
- DW-ES(B) / Fasting condition (Experimental): 625mg
  Interventions: Drug: DW-ES(B)
- Megace / Fed condition (Active Comparator): 800mg
  Interventions: Drug: Megace
- DW-ES(B) / Fed condition (Experimental): 625mg
  Interventions: Drug: DW-ES(B)

INTERVENTIONS:
Drug: Megace — 800mg
  Arms: Megace / Fasting condition; Megace / Fed condition
Drug: DW-ES(B) — 625mg
  Arms: DW-ES(B) / Fasting condition; DW-ES(B) / Fed condition

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics of Daewon DW-ES(B) 625mg/5ml and Megace 800mg/20ml in healthy male volunteers under fasting and fed condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 to 40 years at screening.
* No significant congenital/chronic disease. No symptoms in physical examination.
* Appropriate subjects as determined by past medical history, laboratory tests, serology and urinalysis.
* Be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
* History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety (normal results for safety tests) | 30days
  Adverse events Physical examination, vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr